CLINICAL TRIAL: NCT05601908
Title: Feasibility and Acceptability of a Virtual Reality Relaxation Intervention for Mental Health Staff
Brief Title: A Virtual Reality Relaxation Intervention for Clinical Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMAS15023
Record Dates: First submitted 2022-10-07; First posted 2022-11-01 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Psychological Burnout; Stress, Psychological; Mental Health Burden
Keywords: virtual reality; relaxation; healthcare staff
MeSH Terms: conditions — Burnout, Psychological; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Pre-post-test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR Relaxation (Experimental): a 5-week course of 20-min sessions of VR relaxation
  Interventions: Other: Virtual Reality Relaxation

INTERVENTIONS:
Other: Virtual Reality Relaxation — Participants will undergo a 5-week course of 20-min sessions of VR relaxation. The VR device used will be the Oculus Quest wireless head mounted display (HMD) with two handheld controllers. The HMD and software have been provided by a Germany based company called Magic Horizons. Participants will be asked to wear the HMD and will wear headphones to hear audio. Each session will involve participants experiencing two virtual environments designed to promote relaxation, at least one of which will have a small interactive component to aid engagement. Environments will focus on nature and will be paired with soothing music or guided meditation. For example, scenes might include dolphins dancing underwater, a beach with rock pools, waterfalls, a rainforest, green meadows with flowers, mountains with lakes and/or a sandy desert. Participants will be seated throughout all sessions.
  Other Names: VR relaxation

SUMMARY:
Clinical staff working in mental health services experience high levels of work-related stress, burnout and poor wellbeing. They may work long hours, experience stress directly related to the emotional demands of the role and clinical responsibility, experience physical and psychological burnout and may experience high rates of workplace violence. Poorer wellbeing and high burnout amongst mental health staff has been associated with poorer quality of patient care, higher absenteeism, higher turnover rates, and low morale. Virtual reality (VR) relaxation is a technique whereby experiences of pleasant/ calming environments are accessed via a head mounted display to promote relaxation. The use of VR relaxation facilities in the workplace may provide a pragmatic approach to enabling employees to de-stress, relax and optimise their mental wellbeing and may reduce turnover and improve stress related sick leave across the National Health Service (NHS) workforce.

The research will involve a pre-post-test of 5-weeks of VR relaxation for clinical staff working in mental health settings, including those working in inpatient settings and community teams. The pre-post-test will act as a feasibility trial, the primary aim is thereby to determine whether VR relaxation is feasible and acceptable amongst mental health staff. This feasibility study will evaluate the feasibility and acceptability of a 5-week course of weekly 20-minute sessions of VR relaxation for clinical staff. Feasibility and acceptability measures will be collected and summarised at the end of the trial, including percentage of those recruited who consent to take part, completion and drop-out rates, adverse events, and satisfaction with sessions. The secondary objective is to investigate the impact of the VR relaxation intervention on potential outcome measures for a randomised controlled trial (RCT), including perceived psychological stress, worry, psychological burnout, sleep quality and anxiety. The results from this study will inform a later trial by providing key parameters including recruitment, retention, acceptability, and adherence to the treatment protocol. Additionally, follow-up qualitative interviews will be conducted with staff who engaged in the VR and staff who withdrew, to develop an understanding of attitudes towards the VR relaxation intervention.

DETAILED DESCRIPTION:
Participants: Clinical staff affiliated within South London and Maudsley NHS Trust (SLaM) and working in inpatient and outpatient mental health settings will be recruited. The investigators anticipate recruiting 20-25 participants to the study. This number is based on recruiting a big-enough sample to assess the feasibility of the study and of the resources available.

Procedure: The study will be advertised to prospective participants via a general email to staff via the clinical team leader and email circulars. Posters will be displayed in staff rooms with a request that anyone interested in taking part contact the research team. Staff who display an interest in the study will be emailed a participant information sheet with study details. Once participants have provided online written informed consent to take part, they will be asked to undergo baseline assessments. Baseline assessments will be conducted online using Qualtrics and include: a socio-demographic questionnaire (age, gender, ethnicity, occupation, clinical setting, years of experience, highest level of education), measures of stress, worry, sleep, and burnout. All together, the baseline assessments will take approximately 15 mins to complete.

Following completion of baseline measures, participants will undergo a 5-week course of 20-min sessions of VR relaxation. The VR device used will be the Oculus Quest wireless head mounted display (HMD) with two handheld controllers. The HMD and software have been provided by a Germany based company called Magic Horizons. Participants will be asked to wear the HMD and will wear headphones to hear audio. Each session will involve participants experiencing two virtual environments designed to promote relaxation, at least one of which will have a small interactive component to aid engagement. Environments will focus on nature and will be paired with soothing music or guided meditation. For example, scenes might include dolphins dancing underwater, a beach with rock pools, waterfalls, a rainforest, green meadows with flowers, mountains with lakes and/or a sandy desert. Participants will be seated throughout all sessions. Sessions and assessments will be scheduled in working hours around the participant's clinical duties.

Before and after each session participants will be asked to complete state-measures of psychological wellbeing, and they will be asked to rate satisfaction with each session at session completion and complete a measure of sense of presence. Following completion of the 5-week VR relaxation course, participants will repeat baseline measures of stress, worry, burnout and sleep. Participants who drop out of the intervention will be invited to complete these measures providing they attend a minimum of one VR session. The investigators endeavour to complete pre-assessment measures within one week prior to the first VR session and end of intervention measures within one-week of participants finishing the course of VR. Study measures will be presented using the online survey platform Qualtrics. Participants will enter data independently with a member of the research time present to assist.

Follow-up Qualitative Interviews: Participants will be invited to participate in follow-up interviews and feedback regarding their experiences of the VR relaxation intervention will be sought. It is expected that 20 participants will attend a follow-up interview. Each interview will take approximately 30 minutes to complete. A series of simple open-ended questions will be asked, and participants will answer verbally. The questions will address staff's opinions regarding the acceptability and feasibility of conducting VR relaxation sessions in the workplace, aspects they enjoyed and barriers to implementation. An audio-recording will record responses to these questions when permission has been granted. The qualitative data gained from these questions will be analysed using thematic analysis to understand the main themes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical staff affiliated with South London and Maudsley National Health Service Trust (SLaM) and working in inpatient and outpatient mental health settings
* Aged 18 years or older
* Capacity to provide informed consent.

Exclusion Criteria:

* Staff with a history of epilepsy as there is a possibility that an epileptic episode may be generated by the VR equipment
* Is aged <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of wards and community teams agree to hosting the project and number that do not agree to hosting the VR relaxation project | Through study completion, an average of 22 months
  as assessed via a tally of acceptances and refusals
Number of people who consent to take part | Through study completion, an average of 22 months
  as assessed via a tally of acceptances and refusals
Average adherence to VR relaxation sessions and assessments | Throughout length of participation in the VR trial, 5 weeks
  as assessed via a record of number of VR sessions and number of assessments attended, and number of VR sessions and assessments not attended
Number of Participants With Treatment-Related Adverse Events | Through study completion, an average of 22 months
  as assessed via a tally of all medical effects observed and all medical effects reported by participants
What proportion of participants adhere to the 20-min VR session | Throughout length of participation in the VR trial, 5 weeks
  as assessed via a record of number of VR sessions completed in full (20 minutes) and number of sessions aborted before completion

SECONDARY OUTCOMES:
Change in The Perceived Stress Scale (PSS-10) score | baseline, 5-weeks
  PSS-10 scores range between 0 and 40. Lower scores indicate lower perceived stress. A score of 27 or over is considered high perceived stress.
Change in The Penn State Worry Questionnaire (PSWQ) score | baseline, 5-weeks
  Scores range from 16 to 80 with higher scores indicative of higher levels of trait worry. A score of 52 or above suggested the person is currently having some problems with worry
Change in The Oldenburg Burnout Inventory (OLBI) score | baseline, 5-weeks
  Scores range from 16 to 64 with higher scores indicative of higher burnout. A score of 35 or above has been used to indicate a higher risk of burnout.
Change in The Pittsburgh Sleep Quality Index (PSQI) score | baseline, 5-weeks
  Scores range from 0 to 21 with higher scores indicative of greater difficulty with sleep. A score of 5 or above is considered a significant sleep disturbance.
What proportion of participants successfully complete their personal goal, this will be measured using the Goal Attainment Scaling (GAS) | baseline, 5-weeks
  personalized training goals (e.g. I would like to be able to sleep better) will be operationalised and measured using the GAS and the investigators will record the number of participants who complete their goal and the number who do not

OTHER OUTCOMES:
Change in the Visual Analogue Scale (VAS) 10-point scale score assessing Stress | Before and after each VR session, throughout length of participation in the VR trial, 5 weeks
  Participants asked: 'how stressed do you feel right now?' on a 10-point scale where 0 is not at all and 10 is extremely stressed
Change in the Visual Analogue Scale (VAS) 10-point scale score assessing relaxation | Before and after each VR session, throughout length of participation in the VR trial, 5 weeks
  Participants asked: 'how relaxed do you feel right now?' on a 10-point scale where 0 is not at all and 10 is extremely relaxed
Change in the Visual Analogue Scale (VAS) 10-point scale score assessing tiredness | Before and each each VR session, throughout length of participation in the VR trial, 5 weeks
  Participants asked: 'how sleepy do you feel right now?' on a 10-point scale where 0 is not at all and 10 is extremely sleepy
Change in the Visual Analogue Scale (VAS) 10-point scale score assessing connection to nature | Before and after each VR session, throughout length of participation in the VR trial, 5 weeks
  Participants asked: 'how connected to nature do you feel right now?' on a 10-point scale where 0 is not at all and 10 is extremely connected
Change in The Patient Health Questionnaire-2 (PHDQ-2) score | Before and after each VR session, throughout length of participation in the VR trial, 5 weeks
  Scores range from 0 to 6 with higher scores indicative of lower mood. A score of 3 or above has been used to indicate possible depression.
Change in The Generalized Anxiety Disorder 2-item scale score | before each VR relaxation session throughout length of participation in the VR trial, 5 weeks
  Scores range from 0 to 6 with higher scores indicative of greater generalised anxiety. A score of 3 or above has been used to indicate possible generalized anxiety disorder.
Change in the Visual Analogue Scale (VAS) 10-point scale score assessing sleep quality | before each VR relaxation session throughout length of participation in the VR trial, 5 weeks
  Participants asked to rate how well they have been sleeping in the last week on a 10-point scale where 0 is poorly and 10 is very well
Change in the Slate-Usoh-Steed Sense of Presence Questionnaire (SUS) score modified to this study's VR 'relaxing environment' to measure sense of presence in the virtual environments | after each VR relaxation session throughout length of participation in the VR trial, 5 weeks
  Scores range from 6 to 42 with higher scores indicative of a greater sense of presence in the VR environment.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Riches, PhD, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Trust, London, Greater London, United Kingdom

REFERENCES:
- [Background] Morse G, Salyers MP, Rollins AL, Monroe-DeVita M, Pfahler C. Burnout in mental health services: a review of the problem and its remediation. Adm Policy Ment Health. 2012 Sep;39(5):341-52. doi: 10.1007/s10488-011-0352-1. PMID 21533847
- [Background] d'Ettorre G, Pellicani V. Workplace Violence Toward Mental Healthcare Workers Employed in Psychiatric Wards. Saf Health Work. 2017 Dec;8(4):337-342. doi: 10.1016/j.shaw.2017.01.004. Epub 2017 Feb 6. PMID 29276631
- [Background] Johnson J, Hall LH, Berzins K, Baker J, Melling K, Thompson C. Mental healthcare staff well-being and burnout: A narrative review of trends, causes, implications, and recommendations for future interventions. Int J Ment Health Nurs. 2018 Feb;27(1):20-32. doi: 10.1111/inm.12416. Epub 2017 Dec 15. PMID 29243348
- [Background] Riches S, Azevedo L, Bird L, Pisani S, Valmaggia L. Virtual reality relaxation for the general population: a systematic review. Soc Psychiatry Psychiatr Epidemiol. 2021 Oct;56(10):1707-1727. doi: 10.1007/s00127-021-02110-z. Epub 2021 Jun 13. PMID 34120220
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130